CLINICAL TRIAL: NCT05889221
Title: Multicenter Phase 2 Study of Subcutaneous Isatuximab Plus Bortezomib, Lenalidomide and Dexamethasone in the Treatment of Newly Diagnosed Transplant Ineligible Multiple Myeloma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Collaborators: Sanofi (Industry); Intergroupe Francophone du Myelome (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISASOCUT - IFM2022-05
Record Dates: First submitted 2023-04-25; First posted 2023-06-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Multiple Myeloma; Myeloma Multiple; Myeloma
Keywords: ISATUXIMAB; ISASOCUT; Bortezomib; Lenalidomide; Dexamethasone; VGPR
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Pharmaceutical Preparations; Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination isatuximab SC, lenalidomide, bortezomib and dexamethasone (Experimental)
  Interventions: Other: Drug and medical device

INTERVENTIONS:
Other: Drug and medical device — Isatuximab will be administered in the hospital by an healthcare professional in the periumbilical region at a single site, using an investigational device injector; injection site will be rotated from one administration to the other.

SUMMARY:
Isatuximab was developed on a sub-cutaneous (SC) administration format. SC administration is expected to be more convenient for the patient, with a much shorter duration of administration compared to the currently approved IV route.

The SC Isatuximab RP2D fixed dose was determined at 1400 mg in a phase1b assessing SC Isatuximab in combination with pomalidomide and dexamethasone in RRMM patients. A similar activity and a favorable safety administration profile compared to the IV formulation, was shown in this trial, as expected (Moreau et al, ASH 2021; Quach et al, ASCO 2022). This data should be confirmed in the ongoing IRAKLIA/EFC15951 phase 3 study, that compared in the RRMM, isatuximab plus pomalidomide and dexamethasone IV versus SC. Whether isatuximab SC, fixed 1400 mg dose, will show similar efficacy and safety profile as to anti-CD38Rd+V remains to be demonstrated. The investigators have planned to study the combination of SC isatuximab plus VRd (IsVRd) in patients with NDMM NTE in a phase 2 study across IFM (Intergroupe Francophone du Myeloma) centers in France to compare indirectly this data to the data obtained from studies that have studied this association in that population with the IV isatuximab formulation.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to understand and voluntarily sign an informed consent form
2. Must be able to adhere to the study visit schedule and other protocol requirements
3. Patient able to swallow the various oral treatments
4. Life expectancy > 6 months
5. Subject, male or female, must be at least ≥ 65 years of age
6. Must have a Newly diagnosed Multiple Myeloma requiring therapy (SLiM CRAB criteria) (see appendix 18.2) 6.1. Monoclonal plasma cells in the bone marrow ≥10% or presence of a biopsy proven plasmacytoma 6.2. Revised International Myeloma Working Group diagnostic criteria for multiple myeloma

   Myeloma defining events:
   * Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically: • Hypercalcemia: serum calcium >0.25 mmol/L (>1 mg/dL) higher than the upper limit of normal or >2.75 mmol/L (>11 mg/dL) • Renal insufficiency: creatinine clearance ≤40 mL per min† or serum creatinine ≥177 μmol/L (≥2 mg/dL)

     †Measured or estimated by validated equations
   * Anemia: hemoglobin value of ≥ 20 g/L below the lower limit of normal, or hemoglobin value ≤100 g/L
   * Bone lesions: one or more osteolytic lesions on skeletal radiography, CT, or PET-CT ‡

     * If bone marrow has less than 10% clonal plasma cells, more than one bone lesion is required to distinguish from solitary plasmacytoma with minimal marrow involvement
   * Any one or more of the following biomarkers of malignancy:

     * Clonal bone marrow plasma cell percentage* ≥60%
     * Involved/uninvolved serum free light chain ratio ≥100
     * >1 focal lesion on MRI studies (Each focal lesion must be 5 mm or more in size.)
7. Must have measurable disease as defined by any of the following:

   Serum monoclonal paraprotein (M-protein) level ≥5 g/L or urine M- protein level ≥200 mg/24 hours; or Serum immunoglobulin free light chain ≥100 mg/L and abnormal serum immunoglobulin kappa lambda free light chain ratio (any method)*

   * The same method must be used along the study for a given patient.
8. Must be nontransplant eligible 8.1. Newly diagnosed and not considered candidate for high- dose chemotherapy with SCT. 8.2. Subject must have Charlson comorbidity index ≤1 8.3. ECOG ≤2
9. Adequate bone marrow function, documented within 72 hours and without transfusion 72 hours prior to the first intake of investigational product (C1J1) with no growth factor support (one week), defined as:

   * Absolute neutrophils ≥ 1 x109/L,
   * Untransfused Platelet count ≥ 75 x109/L,
   * Hemoglobin ≥8.5 g/dL.
10. Adequate organ function documented within one week prior to the first intake of investigational product (C1J1) defined as:

    * Serum total bilirubin < 2x upper limit of normal (ULN),
    * Creatinine clearance ≥ 30ml/min calculated with MDRD formula,
    * Serum SGOT/AST or SGPT/ALT < 3x upper limit of normal (ULN).
11. Person affiliated to the French social security system or equivalent
12. A man who is sexually active with a pregnant woman or a woman of childbearing potential must agree to use a barrier method of birth control e.g., condom with spermicidal foam/gel/film/cream/suppository during the study and for at least 5 months after the last dose of treatment, even he has had a vasectomy.
13. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    13.1. Not a female of childbearing potential Or 13.2. A FCBP* who must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours prior to starting study medication and before each cycle of study treatment.

    A FCBP* must understand and agree to continue abstinence from heterosexual intercourse or to use 2 reliable effective methods of contraception (a very effective method and an effective additional method) simultaneously without interruption:

    13.2.1. For at least 28 days before starting experimental treatments, 13.2.2. Throughout the entire duration of experimental treatments, 13.2.3. During dose interruptions, 13.2.4. And for at least 5 months after the last dose of experimental treatments.
14. All patients must understand and accept to comply with the conditions of the Lenalidomide pregnancy prevention plan

Exclusion Criteria :

1. Subject has a diagnosis of primary systemic amyloidosis, monoclonal gammopathy of undetermined significance, or smouldering multiple myeloma.
2. Subject has a diagnosis of Waldenström's disease, or other conditions in which IgM M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions.
3. Subject has prior or current systemic therapy or SCT for multiple myeloma, with the exception of an emergency use of a short course (equivalent of dexamethasone 40 mg/day for a maximum 4 days) of corticosteroids before treatment.
4. Subject has a history of ongoing malignancy (other than multiple myeloma) within 3 years (date of diagnosis of the malignancy) before inclusion in the study treatment (exceptions are malignancies considered cured with minimal risk of recurrence within 3 years, even though the patient receives treatment).
5. Subject has had radiation therapy within 7 days study treatment*

   * unless done for antalgic reason or in case of functional risk for the patient.
6. Subject has had plasmapheresis within 7 days study treatment *

   * unless patient disease is still measurable (inclusion criteria n°6) after the plasmapheresis.
7. Subject is exhibiting clinical signs of meningeal involvement of multiple myeloma.
8. Known to be seropositive for history of human immunodeficiency virus (HIV).
9. Known to have hepatitis B active or uncontrolled infection (positive HBsAg and/or HBV DNA)
10. Known to have hepatitis C active infection (positive HCV RNA and negative anti-HCV)
11. Subject has any clinically significant medical or psychiatric condition or disease (e.g., uncontrolled diabetes, acute diffuse infiltrative pulmonary disease) in the investigator's opinion, would expose the patient to excessive risk or may interfere with compliance or interpretation of the study results.
12. Subject has active systemic infection and severe infections requiring treatment with a parenteral administration of antibiotics.
13. Subject has clinically significant cardiac disease, including:

    * myocardial infarction within 6 months before study treatment, or an unstable or uncontrolled disease/condition related to or affecting cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV)
    * uncontrolled cardiac arrhythmia (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 5 Grade ≥2) or clinically significant ECG abnormalities or LVEF < 40 % 14. Subject has known allergies, hypersensitivity, or intolerance to steroids, mannitol, pregelatinized starch, sodium stearyl fumarate, histidine (as base and hydrochloride salt), arginine hydrochloride, poloxamer 188, sucrose or any of the other components of study intervention that are not amenable to premedication with steroids and H2 blockers or would prohibit further treatment with these agents, monoclonal antibodies or human proteins, or their excipients (refer to respective package inserts or Investigator's Brochure).

      15. Known hypersensitivity, allergy to one of the study product (isatuximab, lenalidomide, bortezomib), dexamethasone, boron or to one of the excipients. Allergy to bandages or adhesives (acrylic).

      16. Acute diffuse infiltrative pneumopathy, pericardial disease 17. Subject has plasma cell leukemia (according to World Health Organization [WHO] criterion: ≥20% of cells in the peripheral blood with an absolute plasma cell count of more than 2 × 109/L) or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).

      18. Subject is known or suspected of not being able to comply with the study protocol (e.g., because of alcoholism, drug dependency, or psychological disorder). Subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol- specified assessments. Subject is taking any prohibited medications.

      19. Subject has had major surgery within 2 weeks before study treatment or has not fully recovered from surgery, excluding surgery related to myeloma.

      20. Subject has received an investigational drug (including investigational vaccines) within 14 days or 5 half-lives of the investigational drug prior to initiation of study intervention, whichever is longer, or used an invasive investigational medical device within 4 weeks before study treatment or is currently enrolled in an interventional investigational study.

      21. Persons referred to in Articles L1121-5 to L1121-8 of the CSP 22. Subject has contraindications to required prophylaxis for deep vein thrombosis and pulmonary embolism.

      23. Incidence of gastrointestinal disease that may significantly alter the absorption of oral drugs.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
VGPR Rate | The primary outcoume will be evaluate up to 8 months after the treatment after treatment has begun.
  The primary outcome is the VGPR rate or better (as best response) using IMWG criteria.

CONTACTS AND LOCATIONS:
Overall Officials: LELEU Xavier, Prof., Principal Investigator — Poitiers University Hospital
Locations (1):
- CHU Poitiers, Poitiers, France